CLINICAL TRIAL: NCT06865664
Title: Phase I Dose Escalation Study of FGFR4 Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults With Recurrent or Refractory Rhabdomyosarcoma
Brief Title: FGFR4 Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults With Recurrent or Refractory Rhabdomyosarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001570; 001570-C
Record Dates: First submitted 2025-03-07; First posted 2025-03-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01-08

CONDITIONS: Rhabdomyosarcoma
Keywords: Sarcoma; Solid Tumor; CAR T Cells; Rhabdomyosarcoma; FGFR4
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma | interventions — fludarabine; Cyclophosphamide; Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Lymphodepleting preparative regimen (fludarabine and cyclophosphamide) followed by infusion of FGFR4-CAR T cells escalation/de-escalation dose levels
  Interventions: Drug: fludarabine; Drug: cyclophosphamide; Drug: cetuximab; Biological: FGFR4-CAR T Cells
- Arm 2 (Experimental): Lymphodepleting preparative regimen (fludarabine and cyclophosphamide) followed by infusion of FGFR4-CAR T cells at the MTD
  Interventions: Drug: fludarabine; Drug: cyclophosphamide; Drug: cetuximab; Biological: FGFR4-CAR T Cells

INTERVENTIONS:
Drug: fludarabine — 30 mg/m2 per day IV on days -5, -4, -3, -2
Drug: cyclophosphamide — 500 mg/m2 per day IV on days -4, -3, -2
Drug: cetuximab — Participants Age >=18 years, based on FDA approved dosing: Loading dose of 400 mg/m2 IV, followed by 250 mg/m2 IV weekly for a total of 4 doses.
  Participants Age <18 years, based on phase I data of cetuximab in children: Dose of 250 mg/m2 IV administered over 1 hour weekly for a total of 4 doses.
Biological: FGFR4-CAR T Cells — Single intravenous (IV) infusion on Day 0

SUMMARY:
Background:

Rhabdomyosarcoma (RMS) is a cancer of soft tissues. It is the most common soft tissue sarcoma seen in children. RMS cancer cells have a protein called FGFR4 on their surface. Researchers want to try a new kind of treatment for RMS: They will collect a person s own T cells, a type of immune cell; then they will change the T cells so they are better able to target the FGFR4 protein and attack RMS tumor cells. The modified T cells are chimeric antigen receptor (CAR) T cells. The treatment in this study is called FGFR4-CAR T cells.

Objective:

To test FGFR4-CAR T cells in children and young adults with RMS.

Eligibility:

People aged 3 to 39 years with RMS. The RMS must have failed to respond or returned after at least 2 rounds of standard treatment.

Design:

Participants will be screened. They will have physical exam, imaging scans, blood tests, and tests of their heart. They may have a tissue sample taken from their tumor.

They will undergo apheresis: Blood will be taken from the body through a catheter. The blood will pass through a machine that separates out the T cells, and the remaining blood will be returned to the body. The collected T cells will be taken to a lab to create FGFR4-CAR T cells.

Once the FGFR4-CART cells are ready, participants can receive these T cells. For 4 days they will receive drugs to prepare their body for the FGFR4-CAR T cells. After this, the modified T cells will be infused into a vein.

Participants will be then monitored closely to watch for any side effects from the CART cells and be followed to see what effect the CART cells have on their tumors. They will have follow-up visits for up to 5 years. Long-term follow-up will be another 10 years.

DETAILED DESCRIPTION:
Background:

* Rhabdomyosarcoma (RMS) is the most common soft tissue sarcoma of childhood with an annual incidence of 4.5 cases per 1 million children and is the third most prevalent extracranial solid tumor of childhood after neuroblastoma and Wilms tumor.
* RMS is divided into two main subtypes, fusion negative (FN-RMS) driven by RAS pathway mutations, and fusion positive rhabdomyosarcoma (FP-RMS) driven by PAX3/PAX7-FOXO1 fusion genes. Patients with low-risk disease have a 5-year overall survival (OS) that approaches 90% and relapse-free survival that has recently improved to 70-80%, albeit with significant toxicity. However, patients with highrisk or recurrent disease have a dismal prognosis (5-year survival <30% or 17% respectively).
* We have previously reported that FGFR4 is expressed universally in RMS, high expression is associated with an adverse outcome, and approximately 10% of FNRMS have activating mutations of FGFR4.
* We recently reported that fusion gene PAX3-FOXO1, the main oncogenic driver of FP-RMS, establishes a super enhancer in the FGFR4 locus, driving its continual high expression.
* FP-RMS patient tumors that harbor the PAX3 fusions are more likely to be metastatic at presentation, relapse despite aggressive therapy, and have very poor survival, underscoring the critical need to develop novel therapeutic strategies for this subset of patients.
* These data indicate that FGFR4 is universally expressed and a driver oncogene in RMS and therefore is a tractable target for immunotherapy.

Objective:

-To estimate the maximum tolerated dose (MTD) of FGFR4-CAR T cells in children and young adults with recurrent or refractory rhabdomyosarcoma following a cyclophosphamide/fludarabine lymphodepletion regimen.

Eligibility:

* Age >= 3 and <= 39 years old
* Weight >= 15 kg
* Confirmed diagnosis of rhabdomyosarcoma
* Relapsed or refractory rhabdomyosarcoma after at least 2 cancer treatment regimens

Design:

* Phase I, dose-escalation scheme will be used at 4 dose levels (DL) (+/- 20%): DL1 (3 x 10^5 transduced T cells/kg); DL2 (1 x 10^6 transduced T cells/kg); DL3: (3 x 10^6 transduced T cells/kg); DL4 (1 x 10^7 transduced T cells/kg), using a standard 3 + 3 dose-escalation design. Dose level -1 (+/- 20%): 1 x 10^5 transduced T cells/kg may be used if toxicity is noted at dose level 1.
* Upon enrollment, apheresis is performed to collect T cells for transduction prior to preparative chemotherapy. Peripheral blood mononuclear cells (PBMC) may be cryopreserved if necessary, prior to initiation of CAR transduction. CAR transduced T cells will be manufactured and cryopreserved prior to administration.
* Participants will receive a standard lymphodepleting preparative regimen of fludarabine (30 mg/m^2/d on Days -5, -4, -3 and -2) and cyclophosphamide (500 mg/m^2/d on Days -4, -3, and -2)
* Day 0: CAR T cell infusion
* Participants will be monitored for toxicity, antitumor response, CAR expansion, and persistence as well as other biologic correlates

ELIGIBILITY:
* INCLUSION CRITERIA
* Histologically confirmed rhabdomyosarcoma by the NCI Department of Pathology.

Note: Since FGFR4 expression is universal in rhabdomyosarcoma, confirmation of FGFR4 expression is not required.

* Relapsed or refractory rhabdomyosarcoma after at least two (2) cancer treatment regimens i.e., participants should have relapsed or progressed after upfront therapy (that includes any systemic chemotherapy with or without local control) as well as at least one salvage therapy (which can be systemic therapy, radiation, or surgery).
* No available alternative curative therapies per standard of care.
* Participants must have measurable disease per RECIST 1.1 or non-measurable disease on imaging.
* Age >= 3 and <= 39 years old.
* Weight >=15 kg.
* Performance status: Karnofsky >= 50% (>= 16 years) or Lansky >= 50% (< 16 years).

Note: Participants who are unable to walk because of paralysis, but who are upright in a wheelchair will be considered ambulatory for calculating the performance score.

* Participants must be willing to accept blood transfusions.
* Adequate organ and marrow function as defined below:

  * Organ: Bone Marrow Function*

    * Laboratory Element: Absolute neutrophil count; Minimum Requirement >= 500/mcL
    * Laboratory Element: Platelets; Minimum Requirement >= 50,000/mcL

      *Transfusion independent (defined as no transfusion in the prior 7 days) for participants without bone marrow involvement. Participants who have bone marrow involvement with tumor are exempt from the platelet requirement and will not be evaluable for hematological toxicities. Participants must not be refractory to transfusions.
  * Organ: Liver Function

    * Laboratory Element: Aspartate aminotransferase (AST); Minimum Requirement <= 5 x upper limit of normal (ULN)
    * Laboratory Element: Alanine aminotransferase (ALT); Minimum Requirement <= 5 x ULN
    * Laboratory Element: Total bilirubin; Minimum Requirement <= 2 x ULN (Note: Participants with Gilbert's syndrome and/or bilirubin elevation due to tumor involvement are allowed to have <= 5 x ULN)

Note: Adult values will be used for calculating hepatic toxicity and determining eligibility

--Organ: Renal Function

* Age: 3 to < 6 years; Maximum serum creatinine (mg/dL): Male - 0.8, Female - 0.8
* Age: 6 to < 10 years; Maximum serum creatinine (mg/dL): Male - 1, Female - 1
* Age: 10 to < 13 years; Maximum serum creatinine (mg/dL): Male - 1.2, Female - 1.2
* Age: 13 to < 16 years; Maximum serum creatinine (mg/dL): Male - 1.5, Female - 1.2
* Age: >= 16 years; Maximum serum creatinine (mg/dL): Male - 1.7, Female - 1.4

OR

* Measured or calculated creatinine clearance or glomerular filtration rate (GFR); Minimum Requirement: >= 60mL/min/1.73 m^2

  --Organ: Cardiac Function
* Laboratory Element: Cardiac status; Minimum Requirement: Cardiac ejection fraction >= 45% or shortening fraction >= 28%, pericardial effusion <= grade 2 as determined by an echocardiogram (ECHO)

  * Organ: Pulmonary Function
* Laboratory Element: Pulmonary status; Minimum Requirement: Pleural effusion <= grade 1; Oxygen (O2) saturation >=92% on room air at rest

  --Organ: Neurological Function
* Laboratory Element: Neurologic status; Minimum Requirement: No acute neurotoxicity greater than grade 2 per CTCAE v.5.0 with the exception of decreased tendon reflex (DTR). Any grade of DTR is eligible.

  * Individuals of child-bearing potential (IOCBP) must agree to use highly effective contraception (hormonal, intrauterine device [IUD], abstinence, surgical sterilization) at the study entry and up to 12 months after the last dose of combined chemotherapy or 6 months after FGFR4-CAR T cells infusion, whichever is later. Individuals who can father children must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) at the study entry and up to 4 months after the last dose of combined chemotherapy or 6 months after FGFR4-CAR T cells infusion, whichever comes later. We also will recommend individuals who can

father children with IOBCP partners ask their partners to be on highly effective birth control (hormonal, IUD, surgical sterilization). Individuals who can father children must not freeze or donate sperm within the same period.

* Nursing participants must be willing to discontinue nursing from study treatment initiation through 4 months after completion of chemotherapy preparative administration or 6 months after FGFR4-CAR T cells infusion, whichever is later.
* Participants with previous central nervous system (CNS) tumor involvement that has been treated and is stable for at least 6 weeks following completion of therapy as evidenced by no requirements for corticosteroids, no evolving neurologic deficits, and no progression

of residual brain abnormalities without specific therapy, are permitted. Participants with asymptomatic subcentemeric CNS lesions are permitted if no immediate radiation or surgery is indicated.

* Participants must be willing to be enrolled into protocol 15C0028 "Follow-Up Evaluation for Gene-Therapy Related Delayed Adverse Events after Participation in Pediatric Oncology Branch Clinical Trials" after 5 years on this trial.
* The ability of participant or parent/guardian to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA

* Prior therapy with the following prior to apheresis:

  * tyrosine kinase inhibitor, targeted agent, or metronomic non-myelosuppressive regimen within <= 1 week
  * systemic chemotherapy within <= 2 weeks
  * antineoplastic antibody therapy, checkpoint inhibitors, or vaccine therapy, within <= 3 weeks or 5 half-lives (whichever is shorter)
  * radiation within <= 3 weeks (<= 6 weeks if CNS or lung fields have been radiated or in case of craniospinal irradiation of radiation of >=50% of bony pelvis and <=12 weeks in case of total body irradiation). Note: There is no time restriction if the volume of bone marrow treated is less than 10% and the participant has measurable/evaluable disease outside the radiation port
  * any investigational agents within <= 4 weeks
  * autologous stem cell infusion following myeloablative therapy within <= 6 weeks
  * genetically modified T cell, NK cell, or dendritic cell therapy within <= 6 weeks
  * allogeneic stem cell transplant/infusion within <=12 weeks or evidence of active graft versus host disease (GVHD)
* Participants receiving more than physiologic dosing of systemic steroids (3 mg/m^2/day of prednisone equivalent).
* History of severe, immediate hypersensitivity reaction attributed to any agents used in the study or in the manufacturing of the cells.
* Second malignancy at any time.
* Primary immunodeficiency.
* Seropositive for human immunodeficiency virus (HIV) antibody.
* Seropositive for hepatitis C (HCV) or positive for Hepatitis B (HBV) surface antigen (HbsAg).
* Pregnancy confirmed with beta-HCG serum or urine pregnancy test performed in IOCBP at screening.
* Uncontrolled intercurrent illness or social situations that would limit compliance with study requirements.

Ages: 3 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Estimate the MTD of FGFR4-CAR T cells in children and young adults with recurrent or refractory rhabdomyosarcoma following a cyclophosphamide/fludarabine lymphodepletion regimen | 28 days
  Estimation of MTD using evaluation of adverse events considered to be a DLT within DLT period as explained in sections Dose Limiting Toxicity (DLT) and Dose Escalation (Arm 1)

SECONDARY OUTCOMES:
Evaluate the feasibility of manufacturing FGFR4-CAR T cells for children and young adults with recurrent or refractory rhabdomyosarcoma | Initiation of manufacturing FGFR4-CAR T cells of the first participant until completion of CART cell manufacturing of the last participant.
  The fraction of participants who can successfully manufacture the targeted dose number meeting the requirements of the certificate of analysis
Evaluate the safety of FGFR4-CAR T cells therapy in children and young adults with recurrent or refractory rhabdomyosarcoma | 6 months
  The frequency of adverse events among treated participants and reporting the results, by maximum grade of event and type of toxicity noted, this will also include a description of the number of participants with CRS at each dose level.
Evaluate progression-free survival | Baseline, Day 30, 3, 6, 9, 12 months after cell infusion, every 3 months after that for year 2, every 12 months for years 3-5.
  PFS will be reported along with 80% and 95% two-sided confidence intervals
Evaluate ORR for those with measurable disease defined as CR + PR according to RECIST 1.1 in children and young adults with rhabdomyosarcoma | Baseline, Day 30, 3, 6, 9, 12 months after cell infusion, every 3 months after that for year 2, every 12 months for years 3-5.
  ORR will be summarized as the fraction of participants with measurable disease who experience a response (PR + CR) by dose level. The best overall response will be based upon the disease assessments recorded during the study visits, and reported by dose level in terms of confirmed CR/PR, unconfirmed CR/PR, SD, or PD

CONTACTS AND LOCATIONS:
Overall Officials: Srivandana Akshintala, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001570-C.html